CLINICAL TRIAL: NCT06360497
Title: The Effect of Mindfulness Meditation and Loving-kindness and Compassion Meditation on Psychological Distress: The Perspective of Reinforcement Sensitivity Theory
Brief Title: The Effect of Mindfulness Meditation and Loving-kindness and Compassion Meditation on Psychological Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202206090070
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: MM Group; LKCM Group; Waitlist Group
Keywords: mindfulness, loving-kindness and compassion
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mindfulness meditation group (Experimental): participants in mindfulness meditation group would receive four weeks mindfulness meditation intervention.
  Interventions: Other: mindfulness meditation intervention and loving-kindness and compassion meditation intervention
- loving-kindness and compassion meditation group (Experimental): participants in loving-kindness and compassion meditation group would receive four weeks loving-kindness and compassion meditation meditation.
  Interventions: Other: mindfulness meditation intervention and loving-kindness and compassion meditation intervention
- waitlist (No Intervention): participants in waitlist receive no intervention

INTERVENTIONS:
Other: mindfulness meditation intervention and loving-kindness and compassion meditation intervention — Interventions were conducted by two teachers separately. Mindfulness meditation group provided the knowledge and practice related with mindfulness, and loving-kindness and compassion meditation group provided knowledge and practice related with loving-kindness and compassion meditation.
  Other Names: waitlist
  Arms: loving-kindness and compassion meditation group; mindfulness meditation group

SUMMARY:
The purpose of the study is to explore the effect of of mindfulness meditation and loving-kindness and compassion meditation on psychological distress (i.e., anxiety, depression, stress), and explore the mechanism from the perspective of reinforcement sensitivity theory.

DETAILED DESCRIPTION:
Participants were randomly assigned to three groups: mindfulness meditation group (MM, n = 51), loving-kindness and compassion meditation group (LKCM, n = 51), and waitlist group (n = 50). Participants in MM group and LKCM group received four weeks intervention, and data was collected before the intervention and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

(1) have not attended structured meditation intervention; (2) have not diagnosed psychiatric diseases; (3) not currently receiving or has never received psychological counseling; (4) not currently taking or has never taken psychotropic medication; (5) age is less than 18.

Exclusion Criteria:

(1) have attended structured meditation intervention; (2) have diagnosed psychiatric diseases; (3) receiving or have received psychological counseling; (4) taking or have taken psychotropic drugs; (5) age is more than 18.

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-10-09 (Actual); Study Completion 2022-10-09 (Actual)

PRIMARY OUTCOMES:
The Depression Anxiety Stress Scale | 2 months
  The scalewas used to measure depression, anxiety, and stress with 21 items. Participants are required to report the degree of conformity scoring from 1 (did not apply to me at all) to 4 (applied to me very much).
The Philadelphia Mindfulness Scale | 2 months
  The scale was used to measure the degree of mindfulness, with 10 items and two dimensions, scoring from 1 (never) to 5 (always).
The Sensitivity to Punishment and Sensitivity to Reward Questionnaire | 2 months
  The scale included 34 items to test the sensitivity to punishment and sensitivity to reward. and participants were asked to respond yes (scoring 1) or no (scoring 0). Summing the scores of the questions was the total score for that dimension.

SECONDARY OUTCOMES:
The Emotional Word Lists | 2 months
  The scale was used to measure emotions, to test the basic effect of interventions. There were 24 emotional words, which constructed two dimensions: positive emotion and negative emotion, scoring from 1 (never) to 5 (always).

CONTACTS AND LOCATIONS:
Locations (1):
- Xianglong Zeng, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT06360497/Prot_SAP_000.pdf